CLINICAL TRIAL: NCT04386941
Title: Holmium Laser Xpeeda Vaporesection Versus Greenlight XPS Vaporization of the Prostate for Benign Prostatic Obstruction: A Randomized Controlled Clinical Study
Brief Title: Greenlight Vaporization vs Xpeeda Vaporesection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thunder Bay Regional Health Research Institute (Other)
Collaborators: Northern Ontario School of Medicine (Other); Thunder Bay Regional Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Hazem Elmansy, Urology Surgeon, Thunder Bay Regional Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: RP-582
Record Dates: First submitted 2020-05-04; First posted 2020-05-13 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Benign Prostatic Hyperplasia; Lower Urinary Tract Symptoms
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms

STUDY DESIGN:
Intervention Model Description: Prospective randomized clinical study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Greenlight XPS Vaporization (Active Comparator): Greenlight 532nm laser photoselective vaporization of the prostate (PVP) is an appealing treatment modality with hemoglobin as tissue target chromophore and relatively short learning curve. The introduction of the Xcelerated Performance System (XPS) 180W in 2010 with the MoXy fibers represents the highest-powered system currently in use for this type of laser. It encourages the adoption of the enucleation principle, making it a real contender to HoLEP in treating large adenomas. Despite the fact that large prostates often require more energy and longer operative time, the XPS system has reduced the operative time and number of fibres required in these situations.
  Interventions: Procedure: Greenlight XPS Vaporization of the Prostate
- Xpeeda Fibre Laser Vaporesection (Active Comparator): Holmium Xpeeda side firing fibre was introduced and it stands apart from other available technologies as a combination of power and efficiency, which minimizes vaporization time. This technology seems to revolutionize utilization of the Holmium power and delivering more energy directly to the tissue, due to its capability of being in contact with the tissue. Moreover, hemostasis would be improved by the pulse reshaping technology with a wider pulse width, activated by a dedicated footswitch. Therefore, the Lumenis Pulse™ 100W will make prostate vaporesection procedures more precise, faster and efficient, with excellent hemostasis. Consequently, bleeding is minimal, tissue is easier to remove and patients can have their catheter removed faster.
  Interventions: Procedure: Xpeeda Fibre Laser Vaporesection of the Prostate

INTERVENTIONS:
Procedure: Xpeeda Fibre Laser Vaporesection of the Prostate — Both interventions are currently used standard of care treatments for the Holmium laser enucleation of the prostate (HoLEP) for patients with bothersome lower urinary tract symptoms (LUTS) secondary to benign prostatic hyperplasia (BPH).
  Holmium Xpeeda side firing fibre was introduced and it stands apart from other available technologies as a combination of power and efficiency, which minimizes vaporization time. This technology seems to revolutionize utilization of the Holmium power and delivering more energy directly to the tissue, due to its capability of being in contact with the tissue.
  Arms: Xpeeda Fibre Laser Vaporesection
Procedure: Greenlight XPS Vaporization of the Prostate — The introduction of the Xcelerated Performance System (XPS) 180W in 2010 with the MoXy fibers represents the highest-powered system currently in use for this type of laser.11 It encourages the adoption of the enucleation principle, making it a real contender to HoLEP in treating large adenomas. Despite the fact that large prostates often require more energy and longer operative time, the XPS system has reduced the operative time and number of fibers required in these situations.
  Arms: Greenlight XPS Vaporization

SUMMARY:
Bothersome lower urinary tract symptoms (LUTS) secondary to benign prostatic hyperplasia (BPH) is a common problem, which impact patients' quality of life. It may lead to serious outcomes, including urinary tract infection, hematuria, bladder stones, urinary retention, hydronephrosis, and rarely renal insufficiency.

Introduction of the Holmium laser enucleation of the prostate (HoLEP) represented a turning point in minimally invasive laser therapy for BPH as it achieves size-independent prostatic cavities similar to simple open prostatectomy with significantly lower perioperative morbidity.

Recently, Holmium Xpeeda side firing fibre was introduced and it stands apart from other available technologies as a combination of power and efficiency, which minimizes vaporization time. This technology seems to revolutionize utilization of the Holmium power and delivering more energy directly to the tissue, due to its capability of being in contact with the tissue.

To date, no outcomes of the new Xpeeda laser fiber have been reported in the literature, which is striving for trials comparing XPS 180W with other competitors such as Holmium vaporesection with the new fiber Xpeeda. Therefore, this study is planned to compare both procedures in improving bothersome LUTS secondary to BPH, and to evaluate safety and cost effectiveness.

DETAILED DESCRIPTION:
Bothersome lower urinary tract symptoms (LUTS) secondary to benign prostatic hyperplasia (BPH) is a common problem, which impact patients' quality of life. It may lead to serious outcomes, including urinary tract infection, hematuria, bladder stones, urinary retention, hydronephrosis, and rarely renal insufficiency. Symptoms of BPH are due to prostatic enlargement, increased smooth muscle tone from the bladder and prostate, and changes in bladder contractility leading to lower urinary tract obstruction, which may cause permanent kidney damage if left untreated.

Introduction of the Holmium laser enucleation of the prostate (HoLEP) represented a turning point in minimally invasive laser therapy for BPH as it achieves size-independent prostatic cavities similar to simple open prostatectomy with significantly lower perioperative morbidity. It has successfully passed the steps of validation through a growing number of well-designed randomized controlled studies to have a high level of evidence for safety and efficacy. The pulsed nature of holmium laser allows the plane of enucleation to be easier to develop and follow and gives superior visibility than the electro-cauterization with less charring of tissue.

HoLEP proved itself as the only endoscopic procedure with superior efficacy compared to the traditional transurethral resection of the prostate (TURP). Furthermore, it is not only safe, effective, size-independent and durable even in patients with coagulopathy, but also more cost-effective than TURP. Meta-analyses have confirmed how well established HoLEP has now become, with a low long-term retreatment rate and the more pronounced improvement in prostate symptoms score and flow rate than after TURP.

Recently, Holmium Xpeeda side firing fibre was introduced and it stands apart from other available technologies as a combination of power and efficiency, which minimizes vaporization time. This technology seems to revolutionize utilization of the Holmium power and delivering more energy directly to the tissue, due to its capability of being in contact with the tissue. Moreover, hemostasis would be improved by the pulse reshaping technology with a wider pulse width, activated by a dedicated footswitch. Therefore, the Lumenis Pulse™ 100W will make prostate vaporesection procedures more precise, faster and efficient, with excellent hemostasis. Consequently, bleeding is minimal, tissue is easier to remove and patients can have their catheter removed faster.

On the other hand, Greenlight 532nm laser photoselective vaporization of the prostate (PVP) is an appealing treatment modality with hemoglobin as tissue target chromophore and relatively short learning curve. The introduction of the Xcelerated Performance System (XPS) 180W in 2010 with the MoXy fibres represents the highest-powered system currently in use for this type of laser. It encourages the adoption of the enucleation principle, making it a real contender to HoLEP in treating large adenomas. Despite the fact that large prostates often require more energy and longer operative time, the XPS system has reduced the operative time and number of fibres required in these situations.

Elmansy et al reported that Greenlight vaporization and Holmium laser ablation of the prostate (HoLAP) are effective surgical treatments for BPH in small to medium prostates. The two techniques have similar functional outcomes and complication rates. Subjective and objective voiding parameters showed significant improvement lasting for up to 3 years, confirming the long lasting, durable effects of each technique.

To date, no outcomes of the new Xpeeda laser fiber have been reported in the literature, which is striving for trials comparing XPS 180W with other competitors such as Holmium vaporesection with the new fiber Xpeeda. Therefore, this study is planned to compare both procedures in improving bothersome LUTS secondary to BPH, and to evaluate safety and cost effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Males over 50 years of age at the time of enrollment
2. Referred to urology for refractory LUTS secondary to BPH
3. Prostate size on preoperative TRUS of 40-80 ml
4. IPSS >15, QOL score ≥3 and Qmax <15 ml/sec
5. Written informed consent to participate in the study
6. Ability to comply with the requirements of the study procedures

Exclusion Criteria:

1. Previous surgical treatment for BPH
2. Presence of bladder stones
3. History of prostate cancer
4. Prostate size > 80 mL or <40 mL
5. History of urethral stenosis or its management
6. Known or suspected neurogenic bladder
7. Participants with active urinary tract infection until appropriately treated
8. Participants with preexisting conditions, which, in the opinion of the investigator, interfere with the conduct of the study.
9. Participants who are uncooperative or cannot follow instructions.
10. Participants who lack the capacity to provide free and informed written consent.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2022-07-10 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
International Prostate Symptom Score (IPSS) | Baseline
  The International Prostate Symptom Score (I-PSS) is based on the answers to seven questions concerning urinary symptoms and one question concerning quality of life. Each question concerning urinary symptoms allows the patient to choose one out of six answers indicating increasing severity of the particular symptom. The answers are assigned points from 0 to 5. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic).
International Prostate Symptom Score (IPSS) | 1 month post-op
  The International Prostate Symptom Score (I-PSS) is based on the answers to seven questions concerning urinary symptoms and one question concerning quality of life. Each question concerning urinary symptoms allows the patient to choose one out of six answers indicating increasing severity of the particular symptom. The answers are assigned points from 0 to 5. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic).
International Prostate Symptom Score (IPSS) | 3 months post-op
  The International Prostate Symptom Score (I-PSS) is based on the answers to seven questions concerning urinary symptoms and one question concerning quality of life. Each question concerning urinary symptoms allows the patient to choose one out of six answers indicating increasing severity of the particular symptom. The answers are assigned points from 0 to 5. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic).
International Prostate Symptom Score (IPSS) | 6 months post-op
  The International Prostate Symptom Score (I-PSS) is based on the answers to seven questions concerning urinary symptoms and one question concerning quality of life. Each question concerning urinary symptoms allows the patient to choose one out of six answers indicating increasing severity of the particular symptom. The answers are assigned points from 0 to 5. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic).
International Prostate Symptom Score (IPSS) | 12 months post-op
  The International Prostate Symptom Score (I-PSS) is based on the answers to seven questions concerning urinary symptoms and one question concerning quality of life. Each question concerning urinary symptoms allows the patient to choose one out of six answers indicating increasing severity of the particular symptom. The answers are assigned points from 0 to 5. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic).
Quality of life (QOL) Due to Urinary Symptoms | Baseline
  One question asking; "If you were to spend the rest of your life with your urinary condition just the way it is now, how would you feel about that? Scored from 0-6 with 0 being "delighted" and 6 being "terrible". Higher the score, the lower the quality of life.
Quality of life (QOL) Due to Urinary Symptoms | 1 month post-op
  One question asking; "If you were to spend the rest of your life with your urinary condition just the way it is now, how would you feel about that? Scored from 0-6 with 0 being "delighted" and 6 being "terrible". Higher the score, the lower the quality of life.
Quality of life (QOL) Due to Urinary Symptoms | 3 months post-op
  One question asking; "If you were to spend the rest of your life with your urinary condition just the way it is now, how would you feel about that? Scored from 0-6 with 0 being "delighted" and 6 being "terrible". Higher the score, the lower the quality of life.
Quality of life (QOL) Due to Urinary Symptoms | 6 months post-op
  One question asking; "If you were to spend the rest of your life with your urinary condition just the way it is now, how would you feel about that? Scored from 0-6 with 0 being "delighted" and 6 being "terrible". Higher the score, the lower the quality of life.
Quality of life (QOL) Due to Urinary Symptoms | 12 months post-op
  One question asking; "If you were to spend the rest of your life with your urinary condition just the way it is now, how would you feel about that? Scored from 0-6 with 0 being "delighted" and 6 being "terrible". Higher the score, the lower the quality of life.
Peak flow rate (Qmax) | Baseline
  Indicates the maximum urine flow rate. In men peak flow rates (Qmax) greater than 15-20 ml/second are considered normal, rates less than 10 ml/second are considered abnormal. This is measured by Uroflowmetry, also called a uroflow test, which measures the flow and force of urine stream during urination.
Peak flow rate (Qmax) | Immediately post-catheter removal
  Indicates the maximum urine flow rate. In men peak flow rates (Qmax) greater than 15-20 ml/second are considered normal, rates less than 10 ml/second are considered abnormal. This is measured by Uroflowmetry, also called a uroflow test, which measures the flow and force of urine stream during urination.
Peak flow rate (Qmax) | 1 month post-op
  Indicates the maximum urine flow rate. In men peak flow rates (Qmax) greater than 15-20 ml/second are considered normal, rates less than 10 ml/second are considered abnormal. This is measured by Uroflowmetry, also called a uroflow test, which measures the flow and force of urine stream during urination.
Peak flow rate (Qmax) | 3 months post-op
  Indicates the maximum urine flow rate. In men peak flow rates (Qmax) greater than 15-20 ml/second are considered normal, rates less than 10 ml/second are considered abnormal. This is measured by Uroflowmetry, also called a uroflow test, which measures the flow and force of urine stream during urination.
Peak flow rate (Qmax) | 6 months post-op
  Indicates the maximum urine flow rate. In men peak flow rates (Qmax) greater than 15-20 ml/second are considered normal, rates less than 10 ml/second are considered abnormal. This is measured by Uroflowmetry, also called a uroflow test, which measures the flow and force of urine stream during urination.
Peak flow rate (Qmax) | 12 months post-op
  Indicates the maximum urine flow rate. In men peak flow rates (Qmax) greater than 15-20 ml/second are considered normal, rates less than 10 ml/second are considered abnormal. This is measured by Uroflowmetry, also called a uroflow test, which measures the flow and force of urine stream during urination.
Post-void residual urine volume (PVR) | Baseline
  The amount of urine retained in the bladder after a voluntary void. Incomplete bladder emptying is diagnosed by postvoid catheterization or ultrasonography showing an elevated residual urine volume. A volume < 50 mL is normal; < 100 mL is usually acceptable in patients > 65 but abnormal in younger patients
Post-void residual urine volume (PVR) | Immediately post-catheter removal
  The amount of urine retained in the bladder after a voluntary void. Incomplete bladder emptying is diagnosed by postvoid catheterization or ultrasonography showing an elevated residual urine volume. A volume < 50 mL is normal; < 100 mL is usually acceptable in patients > 65 but abnormal in younger patients
Post-void residual urine volume (PVR) | 1 month post-op
  The amount of urine retained in the bladder after a voluntary void. Incomplete bladder emptying is diagnosed by postvoid catheterization or ultrasonography showing an elevated residual urine volume. A volume < 50 mL is normal; < 100 mL is usually acceptable in patients > 65 but abnormal in younger patients
Post-void residual urine volume (PVR) | 3 months post-op
  The amount of urine retained in the bladder after a voluntary void. Incomplete bladder emptying is diagnosed by postvoid catheterization or ultrasonography showing an elevated residual urine volume. A volume < 50 mL is normal; < 100 mL is usually acceptable in patients > 65 but abnormal in younger patients
Post-void residual urine volume (PVR) | 6 months post-op
  The amount of urine retained in the bladder after a voluntary void. Incomplete bladder emptying is diagnosed by postvoid catheterization or ultrasonography showing an elevated residual urine volume. A volume < 50 mL is normal; < 100 mL is usually acceptable in patients > 65 but abnormal in younger patients
Post-void residual urine volume (PVR) | 12 months post-op
  The amount of urine retained in the bladder after a voluntary void. Incomplete bladder emptying is diagnosed by postvoid catheterization or ultrasonography showing an elevated residual urine volume. A volume < 50 mL is normal; < 100 mL is usually acceptable in patients > 65 but abnormal in younger patients
Prostate specific antigen (PSA) | Baseline
  The PSA test Measures the level of PSA (protein produced by normal, as well as malignant, cells of the prostate gland) in a blood sample. The normal PSA value is usually stated to be less than 4.0 μg/L. However, because of the fact that benign enlargement of the prostate gland tends to occur as men get older, an age-adjusted scale has been developed: 0-2.5 μg/L = Normal for a man 40-50 yrs; 2.5-3.5 μg/L = Normal for a man 50-60 yrs. For men aged 70 to 79, they suggested a normal serum PSA reference range of 0.0-6.5 ng/mL (0.0-6.5 μg/L).
Prostate specific antigen (PSA) | 3 months post-op
  The PSA test Measures the level of PSA (protein produced by normal, as well as malignant, cells of the prostate gland) in a blood sample. The normal PSA value is usually stated to be less than 4.0 μg/L. However, because of the fact that benign enlargement of the prostate gland tends to occur as men get older, an age-adjusted scale has been developed: 0-2.5 μg/L = Normal for a man 40-50 yrs; 2.5-3.5 μg/L = Normal for a man 50-60 yrs. For men aged 70 to 79, they suggested a normal serum PSA reference range of 0.0-6.5 ng/mL (0.0-6.5 μg/L).
Prostate specific antigen (PSA) | 12 months post-op
  The PSA test Measures the level of PSA (protein produced by normal, as well as malignant, cells of the prostate gland) in a blood sample. The normal PSA value is usually stated to be less than 4.0 μg/L. However, because of the fact that benign enlargement of the prostate gland tends to occur as men get older, an age-adjusted scale has been developed: 0-2.5 μg/L = Normal for a man 40-50 yrs; 2.5-3.5 μg/L = Normal for a man 50-60 yrs. For men aged 70 to 79, they suggested a normal serum PSA reference range of 0.0-6.5 ng/mL (0.0-6.5 μg/L).

SECONDARY OUTCOMES:
Rates of intraoperative adverse events | During surgery
  Rates of complications, such as incidence of bleeding, need for use of monopolar diathermy, duration of surgery, and the operative time/ laser time ratio.
Degree of prostatic size change measured by transrectal ultrasound (TRUS) | Surgery and 3-months post-op
  An ultrasound probe is inserted into the rectum to check the prostate. The probe bounces sound waves off body tissues to make echoes that form a sonogram (computer picture) of the prostate. Sonogram at baseline will be compared to that at 3-months post-op and prostate size measured using online measuring tools.
International index of erectile function-5 (IIEF-5) | Surgery
  The 5-question International Index of Erectile Function (IIEF) Questionnaire is a validated, multidimensional, self-administered investigation that has been found useful in the clinical assessment of erectile dysfunction and treatment outcomes. Questions are scored from 1-5, with lower scores indicating increased levels of erectile dysfunction, while higher scores indicate higher erectile function. The possible scores for the IIEF-5 range from 5 to 25, and erectile dysfunction (ED) is classified into five categories based on the scores: severe (5-7), moderate (8-11), mild to moderate (12-16), mild (17-21), and no ED (22-25).
International index of erectile function-5 (IIEF-5) | 3 months post-op
  The 5-question International Index of Erectile Function (IIEF) Questionnaire is a validated, multidimensional, self-administered investigation that has been found useful in the clinical assessment of erectile dysfunction and treatment outcomes. Questions are scored from 1-5, with lower scores indicating increased levels of erectile dysfunction, while higher scores indicate higher erectile function. The possible scores for the IIEF-5 range from 5 to 25, and erectile dysfunction (ED) is classified into five categories based on the scores: severe (5-7), moderate (8-11), mild to moderate (12-16), mild (17-21), and no ED (22-25).
International index of erectile function-5 (IIEF-5) | 12 months post-op
  The 5-question International Index of Erectile Function (IIEF) Questionnaire is a validated, multidimensional, self-administered investigation that has been found useful in the clinical assessment of erectile dysfunction and treatment outcomes. Questions are scored from 1-5, with lower scores indicating increased levels of erectile dysfunction, while higher scores indicate higher erectile function. The possible scores for the IIEF-5 range from 5 to 25, and erectile dysfunction (ED) is classified into five categories based on the scores: severe (5-7), moderate (8-11), mild to moderate (12-16), mild (17-21), and no ED (22-25).

CONTACTS AND LOCATIONS:
Overall Officials: Hazem Elmansy, MD, Principal Investigator — Thunder Bay Regional Health Sciences Centre
Locations (1):
- Thunder Bay Regional Health Sciences Centre/Thunder Bay Regional Health Research Institute, Thunder Bay, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan to share any participant data with other researchers. Investigator findings may be presented at various national and international conferences, however all data will be de-identified and grouped prior to any dissemination, in an effort to protect participant confidentiality

REFERENCES:
- [Derived] Elmansy H, Zakaria AS, Hodhod A, Shabana W, Ahmad A, Oquendo F, Fathy M, Abbas L, Abdul Hadi R, Kelly R, Kotb A, Shahrour W. Holmium Laser Xpeeda Vaporization vs GreenLight XPS Vaporization of the Prostate for Benign Prostatic Obstruction: 1-Year Results from a Randomized Controlled Clinical Study. J Endourol. 2023 Jun;37(6):706-712. doi: 10.1089/end.2022.0727. Epub 2023 May 22. PMID 37029802